CLINICAL TRIAL: NCT00104390
Title: A Single-blind Phase 1 Study to Assess the Residual Allergenicity of Grass/Rye Pollen Allergoid Using Skin Prick Testing
Brief Title: Assessment of Residual Allergenicity of Grass/Rye Pollen Allergoid Using Skin Prick Testing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GrassMATAMPL101
Record Dates: First submitted 2005-02-28; First posted 2005-03-01 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Type I Hypersensitivity
Keywords: allergy; skin prick test; allergoid; allergenicity; specific immunotherapy
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

INTERVENTIONS:
Biological: Grass MATA MPL

SUMMARY:
The purpose of this study is to evaluate the residual allergenicity of Grass MATA (modified pollen allergen tyrosine adsorbate) by skin prick testing. This is done by a comparison of the wheal response after skin prick testing with aqueous native and modified allergen, modified tyrosine adsorbed allergen and Grass MATA MPL (modified tyrosine adsorbed + MPL).

DETAILED DESCRIPTION:
Grass MATA MPL has been developed to provide pre-seasonal specific immunotherapy for patients with proven type I hypersensitivity to cross reacting grass pollens.

MPL (Monophosphoryl Lipid A), a purified, detoxified glycolipid derived from the cell wall of Salmonella minnesota, is included in the product formulation as an adjuvant to increase the immunogenic effect of the product and to enhance the switch from an allergen-specific TH2 to a TH1-like T cell profile.

The grass pollen extract is modified with glutaraldehyde to produce the active ingredient, an allergoid. This modification reduces the reactivity of the extract with IgE antibody, thus reducing the risk of side effects. However, a simultaneous reduction in other important immunological properties, such as IgG and T cell reactivities, is not seen.

The modification is greater than 75 %, so that only a small amount of unmodified allergen is remaining in the product. The purpose of this study is to assess residual allergenicity of the modified grass/rye pollen in Grass MATA MPL using skin prick testing.

In this skin prick test, the following test products will be compared:

* 7 concentrations of aqueous native allergen
* aqueous modified allergen
* modified tyrosine adsorbed allergen
* Grass MATA MPL (modified tyrosine adsorbed + MPL)

ELIGIBILITY:
Inclusion Criteria:

* Positive skin prick test to grass and rye pollen allergen extract
* Positive skin prick test to positive histamine control
* Negative skin prick test to negative control
* Specific IgE for grass and rye as documented by a RAST or equivalent test
* Females of childbearing potential may enter the study if they have a negative urine pregnancy test and they have been practicing adequate contraception for 3 months prior to the study and continue to do so during the study.

Exclusion Criteria:

* History or presence of acute or subacute atopic dermatitis, chronic dermatitis, urticaria factitia, or urticaria due to physical/chemical influence or any other skin conditions which might interfere with the interpretation of skin prick test results
* Visual inspection of the forearms indicates potential problems with the conduct or interpretation of the skin prick tests; both forearms must be available for testing
* Subject has bronchial asthma or other lower respiratory tract condition (i.e., emphysema, bronchiectasis)
* History or presence of diabetes, cancer or any clinically significant cardiac, metabolic, renal, hepatic, gastrointestinal, dermatologic, venereal, hematologic, neurologic or psychiatric diseases or disorders
* Any clinically significant abnormal laboratory value at Visit 1
* Clinically relevant sensitivity to any common perennial allergen: house dust mites, molds, or epithelia (cat, dog, and horse). Sensitivity will be determined by a skin prick test at Visit 1, a RAST (or equivalent method) at Visit 1, or a documented history of symptoms to perennial allergens. Subjects may be enrolled in the study if they test positive, but have no current or historical symptoms to perennial allergens.
* Clinically relevant sensitivity to any common springtime flowering plant: Birch, Oak, Sycamore, Beech, Ash, and Poplar.

Sensitivity will be determined by a skin prick test at Visit 1, a RAST (or equivalent method) at Visit 1, or a documented history of symptoms to springtime (non-grass/rye) allergens. Subjects may be enrolled in the study if they test positive, but have no current or historical symptoms to these springtime allergens.

* History of auto-immune diseases or rheumatoid diseases
* Subject not allowed to receive adrenalin
* Subject has disorder of tyrosine metabolism (i.e., alcaptonuria, tyrosinemia)
* Subject with diseases interfering with the immune response and have received medication, which could influence the results of this study
* Subject has acute or chronic infection
* History of anaphylaxis, including anaphylactic food allergy, insect venom anaphylaxis, exercise or drug induced anaphylaxis
* History of angioedema
* History of hypersensitivity to the excipients of the study medication
* History of immunotherapy with grass allergen extracts
* Current therapy with ß-blockers
* Currently receiving anti-allergy medication or other drugs with an antihistaminic activity
* Subject has a positive drugs of abuse screen at Visit 1
* Subject participated in a clinical trial with an investigational drug within the last 3 months
* Subject cannot communicate reliably with the Investigator or is not likely to cooperate with the requirements of the study
* Subject is pregnant or lactating
* Subject received treatment with a preparation containing MPL during the past 12 months
* Use of prohibited medications or inadequate washout periods prior to screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14
Dates: Start 2005-03; Study Completion 2005-04

PRIMARY OUTCOMES:
to assess the allergenicity of the modified grass/rye pollen allergoid using skin prick testing

SECONDARY OUTCOMES:
evaluation for potential late phase reactions
adverse events
clinical labs
vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Noonan, MD, Principal Investigator — Allergy Associates Research Center
Locations (1):
- Allergy Associates Research Center, Portland, Oregon, United States